CLINICAL TRIAL: NCT03479983
Title: A Randomized, Placebo-Controlled, Parallel-Group, Double-Blind Study of Phyllanthus Emblica L. Fruit Extract (AMX160) in Patients With Hypercholesterolemia
Brief Title: Effect of Indian Gooseberry Extract (AMX160) in Hypercholesterolemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arjuna Natural Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AN-06ASE 0717H4-YSM01
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Hypercholesterolemia
Keywords: Indian gooseberry; Total cholesterol; Triglycerides
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMX160 (Experimental): 500 mg (one capsule) x 2 times daily for 90 days
  Interventions: Dietary Supplement: AMX160
- Placebo (Placebo Comparator): 500mg (one capsule) x 2 times daily for 90 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AMX160 — 500 mg Phyllanthus emblica L. fresh fruit extract capsules
  Other Names: Phyllanthus emblica L.; Indian Gooseberry; Emblica officinalis
  Arms: AMX160
Dietary Supplement: Placebo — 500 mg roasted rice powder in visually identical capsules
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy of a fresh fruit extract of Indian Gooseberry (AMX160) for the attenuation of increased blood cholesterol, LDL cholesterol and triglycerides in patients with hypercholesterolemia.

DETAILED DESCRIPTION:
Phyllanthus emblica L. fruit (Emblica officinalis) has potent antioxidant properties. Animal studies indicate that flavanoids from E. officinalis effectively reduced lipid levels in serum and tissues and had a significant inhibitory effect on hepatic hydroxymethylglutaryl-coenzyme A reductase activity.

The primary aim of this study is to determine whether Phyllanthus emblica L. fruit extract AMX160 is an effective treatment for hypercholesterolemia patients as compared to placebo. The investigators hypothesize that Phyllanthus emblica L. fruit extract AMX160 will significantly lower the total cholesterol as compared to placebo in patients with Hypercholesterolemia. A total of 132 patients including males and females with hypercholesterolemia will be assigned at random to one of the two investigational products. The study is expected to have a treatment duration of 90 ± 10 days and a total duration of 118 days including 14 days of grace period and 14 days of screening period per patient.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males and females aged 18 to 65 years with hypercholesterolemia symptoms: blood Triglycerides, >200 mg/dL, blood cholesterol >200 mg/dL, blood LDL cholesterol >130 mg/dL

Other requirements for inclusion in the study are:

2. Moderate-intensity physical activity (less than 150 minutes or less than 75 minutes of vigorous-intensity physical activity throughout the week) 3. No medication taken for management of hypercholesterolemia during last 4 weeks.

4. Ability to understand and provide signed informed consent. 5. Ability to participate in the study.

Exclusion Criteria:

1. Uncontrolled cardiovascular disease or advanced atherosclerosis (e.g. history of stroke, myocardial infarction, life- threatening arrhythmia, or coronary revascularization within the preceding 6 months; unstable angina; congestive heart failure; known or suspected clinically significant valvular heart disease or uncontrolled hypertension (>160/100 mm of Hg or use of antihypertensive medications, dose of which is not stable in the last one month)
2. Very high triglyceride levels i.e. > 500 mg/dL
3. Diabetes (Fasting Blood Sugar>150 mg/dL), using insulin, glitazones , another hypoglycemic dose of which is not stable in last one month
4. Pregnancy, lactation and female patients not using acceptable contraceptive measures (double barrier methods, oral or injectable hormonal contraceptives or surgical sterilization)
5. Hepatic impairment (Alanine transaminase or Aspartate transaminase levels > 3.0 mg/dl Upper Limit of Normal (ULN)) or renal impairment (serum creatinine≥ 2.0 mg/dl)
6. Severe systemic illness and in the opinion of the investigator would be noncompliant with the visit schedule or study procedures
7. Known history of hypersensitivity to Indian Gooseberry or any product containing Indian Gooseberry extract
8. Patients with history of alcohol intake (For females >3 drinks / day or >7 drinks / week. For Males >4 drinks/ day or > 14 drinks / week).
9. Patients taking any narcotics and prohibited substances.
10. Serious concurrent illness or malignancy.
11. Agreements of participation in another clinical trial in the past 3 months
12. Two of the following risk factors:

    1. Cigarette smoking (Current / Previous smoker < 1 yr)
    2. Hypertension (BP >140/90 mmHg or on antihypertensive medication)
    3. Low HDL cholesterol (<40 mg/dL)
    4. Family history of premature CHD (CHD in male first degree relative <55 years; CHD in female first degree relative <65 years).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Change in Total Cholesterol | Baseline, Day 45 & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.

SECONDARY OUTCOMES:
Change in Triglycerides | Baseline, Day 45 & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.
Change in Low Density Lipoprotein Cholesterol | Baseline, Day 45 & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.
Change in High Density Lipoprotein Cholesterol | Baseline, Day 45 & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.
Change in Very Low Density Lipoprotein Cholesterol | Baseline, Day 45 & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.
Change in Triglyceride /High Density Lipoprotein Cholesterol ratio | Baseline, Day 45 & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.
Change in Apolipoprotein A-1 | Baseline & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.
Change in Apolipoprotein B | Baseline & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.
Change in Apolipoprotein B/Apolipoprotein A-1 Ratio | Baseline & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.
Change in hydroxymethylglutaryl-coenzyme A | Baseline & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.
Change in Coenzyme Q10 | Baseline & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.
Change in Atherogenic index of Plasma | Baseline & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.
Change in Adult Treatment Panel III goal (Triglyceride < 150 mg/dL, LDL < 100 mg/dL, HDL > 40) | Baseline & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.

OTHER OUTCOMES:
Change in Thyroid-stimulating hormone | Baseline & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.
Change in Homocysteine | Baseline & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.
Change in High Sensitivity C-Reactive Protein | Baseline & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.
Change in Global Physical Activity Questionnaire | Baseline & Day 90
  The change over time from the baseline to end of treatment, both within and between the group.

CONTACTS AND LOCATIONS:
Overall Officials: Hamayak Sisakian, MD, Principal Investigator — Yerevan State Medical University, Armenia
Locations (1):
- Clinic of General and Invasive Cardiology University Hospital 1, YSMU, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing can be carried out through a proper research proposal to the scientific review board of Arjuna Natural Ltd except in cases where Arjuna Natural Ltd. has no legal authority because the product has been out-licensed to another company or there is no feasible means to anonymise the data and redact personally identifiable information without compromising the privacy and confidentiality of research participants.